CLINICAL TRIAL: NCT04586725
Title: The Effect of Encouragement on Six Minute Walk Test Performance in Patients With Intermittent Claudication
Brief Title: Effect of Encouragement on Six Minute Walk Test Performance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Central Lancashire (Other)
Collaborators: Coventry University (Other); University of Hull (Other); University of Salford (Other)
Responsible Party: Principal Investigator, Stefan Birkett, Lecturer In Exercise Science, University of Central Lancashire
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: UCentalLancashire2
Record Dates: First submitted 2020-10-07; First posted 2020-10-14 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-07

CONDITIONS: Intermittent Claudication
MeSH Terms: conditions — Intermittent Claudication

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will be blinded to the level of encouragement they will receive during the tests
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Encouragement every minute (Active Comparator): Patients will be randomised to six tests at one week apart
  Interventions: Other: Encouragement a one minute intervals; Other: Encouragement a two minute intervals
- Encouragement every two minutes (Active Comparator): Patients will be randomised to six tests at one week apart
  Interventions: Other: Encouragement a one minute intervals; Other: Encouragement a two minute intervals

INTERVENTIONS:
Other: Encouragement a one minute intervals — Patients will perform the six exercise tests with encouragement at one minute intervals
Other: Encouragement a two minute intervals — Patients will perform the six exercise tests with encouragement at two minute intervals

SUMMARY:
Peripheral artery disease (PAD) is characterised by a build up of fatty plaque in the arteries in the lower limbs, resulting in a reduction of blow flow to the muscles. Globally, it is estimated that 236 million people are living with PAD. A classic symptom of PAD is intermittent claudication (IC) which is characterised by muscle cramps in the lower limbs, typically brought on by exercise and relieved at rest. Exercise is recommended at first line treatment for IC. However to assess IC symptoms in response to an exercise study, maximal walking capacity (the furthest they can walk before it becomes too painful to walk) is typically the main measure. A patients walking capacity is assessed by a number of exercise testing protocols including the six-minute walk test (6MWT), where patients walk for six minutes with the aim to walk as far as they can in the time allotted. Patient encouragement has been shown to improve walking performance by as much as 30 meters in heart failure and respiratory disease populations. However the effect of encouragement on walking performance in people with IC is yet to be studied.

DETAILED DESCRIPTION:
Peripheral artery disease (PAD) is characterised by atherosclerotic lesions of the arteries in the lower limbs, resulting in a reduction of blow flow (Hiatt, 2001). Globally, it is estimated that 236 million people are living with PAD, with the number of cases increasing by 24% from 2000 to 2010. A classic symptom of PAD is intermittent claudication (IC), characterised by ischemic muscle pain precipitated by exertion and relieved by rest. IC is associated with various comorbidities such as diabetes mellitus, hypertension and dyslipidaemia as well as reductions in physical function, quality of life, and balance. National and international guidelines recommend supervised exercise therapy as first line treatment for patients with IC.

To assess IC impairment in response to an exercise intervention, maximal walking capacity is typically the primary outcome in randomised controlled trials (RCT's). This involves a patient walking for as long as possible until ischemic leg symptoms, fatigue or other symptoms prevent them from continuing. This is assessed by a number of exercise testing protocols including the six-minute walk test (6MWT). The American Thoracic Society provide guidelines for performing a standardised 6MWT including verbal phrases that are conducted every minute. Conversely, Montgomery and Gardner suggest encouragement every two minutes. Encouragement has been shown to significantly affect walking performance by as much as 30 meters in heart failure and respiratory disease populations. However the effect of encouragement on walking performance in people with IC is yet to be investigated.

ELIGIBILITY:
Inclusion Criteria:

1. >18 years old
2. Resting ankle brachial pressure index (ABPI) <0.9 or a reduction of ≥ 20 mmHg following exercise testing (per site protocol)
3. Able to walk unaided
4. English speaking and able to follow exercise instructions
5. Able to provide informed consent

Exclusion Criteria:

1. Those who have critical limb threatening ischaemia (rest pain and/or tissue loss)
2. Unable to provide consent
3. Those presenting with any significant comorbidities or contraindications to exercise testing or training in accordance to the American College of Sports Medicine
4. Uncontrolled or symptom limiting coronary heart or pulmonary disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Maximal walking distance (MWD) | 6 weeks
  Metres walked during the tests

SECONDARY OUTCOMES:
Learning effect metres walked | 6 weeks
  To see if a learning effect exists between tests

IPD SHARING:
Plan to Share IPD: No